CLINICAL TRIAL: NCT07299812
Title: BRAVE-HEART: Breast Cancer Radiotherapy Using Active Breathing Coordinator to aVoid Exposure of HEART
Acronym: BRAVE-HEART
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Elisabetta Bonzano, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: BRAVE-HEART
Record Dates: First submitted 2025-11-14; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Radiotherapy
Keywords: Breast cancer; Radiation therapy; Deep inspiration breath hold (DIBH); Cardiac dose; Heart sparing; Active Breathing Coordinator (ABC); Dosimetric analysis; Elderly breast cancer; Simultaneous Integrated Boost (SIB); Hypofractionated radiotherapy; Ultrahypofractionated radiotherapy; Conventional fractionation; Three-dimensional conformal radiotherapy (3D-CRT); Intensity-modulated radiotherapy (IMRT); Volumetric modulated arc therapy (VMAT); Cardiotoxicity; Breast radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Breast cancer patients treated with radiotherapy: Single ambispective observational cohort of patients with breast cancer undergoing radiotherapy according to institutional clinical practice. Within this cohort, eligible patients are treated with the Active Breathing Coordinator-assisted Deep Inspiration Breath Hold (DIBH) technique. Free-breathing treatment plans or patients treated in free-breathing conditions are used as dosimetric references to estimate the reduction in radiation doses to the heart and cardiac substructures achievable with DIBH. Assignment to DIBH or free-breathing conditions is non-randomized and based on clinical suitability and patient cooperation
  Interventions: Radiation: Breast Radiotherapy with or without Deep Inspiration Breath Hold (DIBH)

INTERVENTIONS:
Radiation: Breast Radiotherapy with or without Deep Inspiration Breath Hold (DIBH) — Observational study of breast cancer patients treated with radiotherapy delivered using the Active Breathing Coordinator (ABC) system during Deep Inspiration Breath Hold (DIBH), as implemented in standard clinical practice. Free-breathing treatment plans or patients treated in free-breathing conditions are used as dosimetric references to estimate the reduction in radiation doses to the heart and cardiac substructures achievable with DIBH.

SUMMARY:
The BRAVE-HEART trial is an ambispective, observational, non-randomized study conducted at Fondazione IRCCS (Istituto di Ricovero e Cura a Carattere Scientifico) Policlinico San Matteo (Pavia, Italy). It aims to document and quantify the cardiac dose reduction achievable with breast radiotherapy performed in Deep Inspiration Breath Hold (DIBH) using the Active Breathing Coordinator (ABC) system. Dosimetric parameters from DIBH treatments are evaluated, with free-breathing treatment plans and data from patients treated under free-breathing conditions used as reference. Secondary analyses include treatment reproducibility, comparison of radiotherapy techniques and fractionation schedules, impact of the simultaneous integrated boost (SIB), and assessment of acute and late toxicity during follow-up.

DETAILED DESCRIPTION:
The BRAVE-HEART study is an ambispective, observational, non-randomized, single-center study conducted at Fondazione IRCCS Policlinico San Matteo (Pavia, Italy). The purpose of the study is to document and quantify the heart-sparing effect of breast radiotherapy delivered with Deep Inspiration Breath Hold (DIBH) assisted by the Active Breathing Coordinator (ABC), as implemented in routine clinical practice.

The study includes patients with stage I-III breast carcinoma undergoing radiotherapy according to institutional standards, most commonly after conservative or radical surgery. Radiotherapy is delivered using three-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated/volumetric modulated arc therapy (IMRT/VMAT) techniques, with conventional, hypofractionated, or ultrahypofractionated regimens, with or without a simultaneous integrated boost (SIB) to the tumor bed.

Eligibility for ABC-assisted DIBH is assessed at CT simulation. Patients unable to perform or maintain the breath-hold maneuver are treated under free-breathing conditions. Free-breathing treatment plans and data from patients treated under free-breathing conditions are used as dosimetric references to quantify the magnitude of cardiac dose reduction achievable with ABC-assisted DIBH.

The primary objective is to assess the reduction in radiation dose delivered to the heart and its substructures, particularly the left anterior descending coronary artery (LAD), when radiotherapy is performed with ABC-assisted DIBH. Secondary objectives include evaluating treatment reproducibility and the feasibility of ABC-DIBH in daily practice, comparing dosimetric parameters among different radiotherapy techniques (3D-CRT vs VMAT/IMRT), describing the impact of different fractionation schemes (conventional, hypofractionated, and ultrahypofractionated) and SIB on organs-at-risk exposure, and collecting data on acute and late toxicity during follow-up.

The study aims to provide real-world evidence on the effectiveness, reproducibility, and clinical applicability of ABC-assisted DIBH for cardiac sparing in breast cancer radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-III breast carcinoma with an indication for radiotherapy
* Invasive carcinoma or ductal carcinoma in situ (DCIS)
* Radiotherapy delivered using three-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated/volumetric modulated arc therapy (IMRT/VMAT) techniques
* Ability to actively cooperate in using the Active Breathing Coordinator (ABC) system for Deep Inspiration Breath Hold (DIBH), or treated under free-breathing conditions when DIBH is not feasible
* Age ≥18 years
* Ability to provide written informed consent for the anonymous use of data for research purposes

Exclusion Criteria:

* Severe health problems or profound hearing loss
* Severe respiratory or cardiovascular conditions in the medical history that contraindicate radiotherapy
* Inability to provide written informed consent for the anonymous use of data for research purposes
* Absolute contraindications to radiotherapy (e.g., pregnancy, or inability to maintain the correct treatment position)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambispective cohort of patients with stage I-III breast carcinoma treated with radiotherapy at Fondazione IRCCS Policlinico San Matteo. Radiotherapy may include whole or partial breast or chest wall, with or without nodal irradiation, delivered with 3D-CRT or IMRT/VMAT. The Active Breathing Coordinator (ABC) system is used for DIBH when feasible; patients unable to perform DIBH are treated under free-breathing conditions. Different fractionation schedules and SIB may be used according to clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in mean heart dose (Dmean, Gy) with ABC-assisted DIBH | At baseline RT planning (Day 1)
  Measurement of mean heart dose (Dmean, Gy) in breast cancer patients treated with radiotherapy using ABC-assisted Deep Inspiration Breath Hold (DIBH). Dosimetric comparisons are performed using corresponding free-breathing treatment plans or data from patients treated under free-breathing conditions. All Dmean (Gy) values are derived from the dose-volume histogram (DVH) to evaluate changes in cardiac radiation exposure associated with DIBH.
Change in mean dose (Dmean, Gy) to cardiac substructures with ABC-assisted DIBH | At baseline RT planning (Day 1)
  Change in mean dose (Dmean, Gy) to predefined cardiac substructures (left anterior descending coronary artery, left ventricle) between DIBH and corresponding free-breathing plans or data from patients treated under free-breathing conditions. All Dmean (Gy) values are derived from the dose-volume histogram (DVH).
Change in maximum dose (Dmax, Gy) to cardiac substructures with ABC-assisted DIBH | At baseline RT planning (Day 1)
  Change in maximum dose (Dmax, Gy) to predefined cardiac substructures (left anterior descending coronary artery, left ventricle) between DIBH and corresponding free-breathing plans or data from patients treated under free-breathing conditions. All Dmax (Gy) values are derived from the dose-volume histogram (DVH).

SECONDARY OUTCOMES:
Treatment setup reproducibility using ABC-DIBH | At treatment completion (within 1 week of last fraction)
  Assessment of setup accuracy in patients receiving left-sided breast cancer radiotherapy using deep inspiration breath-hold (DIBH), measured as translational setup shifts (mm) on daily verification imaging.
Dosimetric comparison between 3D conformal radiotherapy and VMAT/IMRT plans | At baseline RT planning (Day 1)
  Analysis of dose-volume histogram (DVH) parameters for target volumes and organs at risk to compare 3D-CRT and VMAT/IMRT techniques in patients treated with breast radiotherapy.
Impact of different fractionation schemes on cardiac and lung doses | At baseline RT planning (Day 1)
  Descriptive analysis of dosimetric parameters (heart Dmean, LAD Dmax/Dmean, ipsilateral lung Dmean, Gy) according to the fractionation schedule adopted (conventional, hypofractionated, and ultrahypofractionated regimens), in patients treated with radiotherapy using DIBH or free-breathing.
Radiotherapy-related toxicity (acute) | 90 days after radiotherapy
  Collection and grading of acute toxicity during radiotherapy according to institutional or CTCAE criteria, in patients treated with DIBH or free-breathing.
Radiotherapy-related toxicity (late) | 12-month follow-up
  Collection and grading of late toxicity during follow-up, according to institutional or CTCAE criteria, in patients treated with DIBH or free-breathing.
Identification of dosimetric cut-offs for cardiac sparing | At baseline RT planning (Day 1)
  Exploratory analysis to identify candidate dose (Gy) thresholds for the heart and left anterior descending coronary artery (LAD), based on the distribution of dose-volume histogram (DVH) parameters within the study cohort. These exploratory dosimetric cut-offs will be considered as potential reference values for cardiac sparing in future studies.
Change in dosimetric parameters with the use of a simultaneous integrated boost (SIB) | At baseline RT planning (Day 1)
  Assessment of changes in predefined dosimetric parameters associated with the use of a simultaneous integrated boost (SIB) in breast radiotherapy delivered according to institutional clinical practice, including treatments performed with ABC-assisted Deep Inspiration Breath Hold (DIBH) or under free-breathing conditions. The analysis includes target coverage metrics (PTV) and organ-at-risk dose metrics (heart and lung; Gy). Comparisons are performed between treatment plans generated with and without SIB within the study cohort. All values are derived from the dose-volume histogram (DVH).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy